CLINICAL TRIAL: NCT04925856
Title: Immunomonitoring of Breast Cancer Patients During Systemic Treatment
Acronym: IMMUNE CAPTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02195-52
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: immune response; blood samples
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): 4 différents cohorts:
  * Paclitaxel cohort (N=30)
  * Epirubicine - cyclophosphamide cohort (N=30)
  * Eribuline cohort (N=30)
  * Palbociclib (N=20) ou Abemaciclib (N=20) ou Ribociclib cohort (N=21)
  Study diagram :
  * Inclusion and screening visite
  * Visit 1: J1C1
  * Visit 2 : J8C1 to Paclitaxel cohort / Epirubicine - cyclophosphamide cohort / Eribuline cohort and J15C1 to Palbociclib ou Abemaciclib ou Ribociclib cohort
  * Visit 3 :J21C1
  * Visit 4 : J8C3 to Paclitaxel cohort / Epirubicine - cyclophosphamide cohort / Eribuline cohort and J15C3 to Palbociclib ou Abemaciclib ou Ribociclib cohort
  During these visits, we collect, before the start of treatment administration ;
  * Vital signs,
  * Concomitant treatments,
  * Blood sample:
    * 1 heparinized tube (4 mL) for collection of plasma and storage
    * 1 heparinized tube (4 mL) for immunophenotyping,
    * 4 EDTA tubes (4 x 10 mL) for collecting white blood cells (PBMC) for cryopreservation.
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — •Blood sample:
  * 1 heparinized tube (4 mL) for collection of plasma and storage
  * 1 heparinized tube (4 mL) for immunophenotyping,
  * 4 EDTA tubes (4 x 10 mL) for collecting white blood cells (PBMC) for cryopreservation.

SUMMARY:
This study aims to constitute a most complete biological collection for patients treated for localized or metastatic breast cancer (in different cohorts depending on the type of systemic treatment received), in order to describe the basal immune response of patients treated for a breast cancer according to the stage of the disease, but above all to study how the different systemic treatments used in the management of breast cancer modulate this immune response.

DETAILED DESCRIPTION:
The main objective of this study is to describe, depending on the type of systemic treatment received, the blood immune response before treatment and its evolution under treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Woman aged between 18 and 85.
2. Patient with histologically proven infiltrating breast cancer.
3. Triple negative breast cancer or RH + / HER2- (OR and RP <10% and HER2 negative (0 or 1+ in IHC or 2+ in IHC and FISH negative)
4. Patient receiving treatment corresponding to one of these cohorts:

   * In a metastatic situation with establishment of treatment with Paclitaxel regardless of the treatment line
   * In a metastatic situation with establishment of treatment with Epirubicin - cyclophosphamide (EC) regardless of the treatment line
   * In a metastatic situation with establishment of treatment with Eribulin regardless of the line of treatment
   * In a 1st line metastatic situation with initiation of treatment with Palbociclib or Abemaciclib, or Ribociclib in combination with hormone therapy (aromatase inhibitor)
5. Patient who signed the informed consent for the study.
6. Patient fit and able to adhere to protocol for the duration of the study, including visits, scheduled specimens and follow-up.
7. Patient affiliated to the social security system.

Exclusion Criteria:

1. Patient unable to understand, read and / or sign informed consent.
2. Presence of cerebral or meningeal metastasis
3. Current or previous use of an immunosuppressive drug in the 14 days preceding inclusion (except intranasal corticosteroids, systemic corticosteroids at physiological doses not exceeding 10 mg per day of prednisone or its equivalent, corticosteroids for antiemetic purposes, corticosteroids used as premedication for hypersensitivity reactions (injected CT scan, taxanes, etc.)
4. Patient participating in another research that may modify the systemic treatment administered in the framework of the cohort in which she will be included.
5. Pregnant or breastfeeding woman.
6. HIV and / or HBV and / or HCV serology positive.
7. Life expectancy estimated at less than 3 months.
8. Patient's refusal.
9. Person benefiting from a protection system for adults (including tutorship and curatorship).
10. Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2030-05-26 (Estimated); Study Completion 2030-05-26 (Estimated)

PRIMARY OUTCOMES:
blood immune response blood immune response blood immune response | 24 months
  realization of a plasma library, immunophenotyping and a PBMC bank
  realization of a plasma library, immunophenotyping and a PBMC bank
  realization of a plasma library, immunophenotyping and a PBMC bank
  realization of a plasma library, immunophenotyping and a PBMC bank
  realization of a plasma library, immunophenotyping and a PBMC bank

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain LADOIRE, PU-PH, Principal Investigator — Centre Georges François Leclerc
Locations (2):
- France (2):
  - CHRU Jean Minjoz, Besançon
  - Centre Georges Francois Leclerc, Dijon